CLINICAL TRIAL: NCT07357168
Title: Effect of Electromagnetic Field Therapy Versus Aerobic Exercise on Prostatic Function in Elderly With Benign Prostatic Hyperplasia
Brief Title: Electromagnetic Field Therapy Versus Aerobic Exercise on Prostatic Function in Elderly With Benign Prostatic Hyperplasia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, El-Sayed Essam, El-Sayed Essam, Cairo University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: (P.T.REC/012/004895)
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Benign Prostate Enlargement
Keywords: electromagnetic field, aerobic exercise
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: The design of the study was randomized controlled trial (RCT), pre test, post test assessment.This study was carried out on seventy five male elderly patients diagnosed with benign prostatic hyperplasia. Their age ranged from 60 to 75 years old.
  The patients of this study were randomly assigned into three equal groups (n= 25):
  Group A (Study group): received pulsed electromagnetic field therapy in addition to medcial treatment program.
  Group B (Study group): received aerobic exercise training in addition to medical treatment program.
  Group C (Control group): received the medical treatment program only.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pulsed electro magnetic field therapy (Active Comparator): It was applied for patients in the study group (A) only for 25 minutes per session, three times per week, for 12 consecutive weeks.
  Interventions: Device: pulsed electromagnetic field
- aerobic exercise training (Active Comparator): It was applied for patients in the study group (B) only. Each session started with 10 minutes of warm-up, followed by treadmill walking for up to 20-30 minutes and ended with a phase of 10 minutes of cool-down.
  Interventions: Device: Treadmill machine
- Routine medical treatment (Other): It was conducted for the three groups (A), (B), and (C).
  Interventions: Device: pulsed electromagnetic field; Device: Treadmill machine

INTERVENTIONS:
Device: pulsed electromagnetic field — It was applied for all patient in the study group (A) only for 25 minutes per session, three times per week, for 12 consecutive weeks
  Arms: Pulsed electro magnetic field therapy; Routine medical treatment
Device: Treadmill machine — was applied for all patients in the study group (B) only. Each session started with 10 minutes of warm-up (dynamic stretching mainly of the lower limbs, ten right and left hip rotations, and ten arm rotations forward and backward), followed by treadmill walking for up to 20-30 minutes and ended with a phase of 10 minutes of cool-down. During the training, the patient was asked to correct the posture during walking with verbal instructions.
  Arms: Routine medical treatment; aerobic exercise training

SUMMARY:
This study will be carried out on seventy five elderly patients with benign prostatic hyperplasia. Their age will range from 60 to 75 years old. They will be recruited from Hoda Talaat Harb geriatric care center, Helwan governorate, Egypt. The aim of this study to investigate the effect of Electromagnetic field versus aerobic exercise on benign prostatic hyperplasia. Benign prostatic hyperplasia is a nonmalignant enlargement of the prostate gland and refers to the stromal and glandular epithelial hyperplasia that occurs in the transition zone of the prostate Clinically, the condition manifests with lower urinary tract symptoms (LUTS) consisting of obstructive (weak urination stream, incomplete bladder emptying, hesitancy) and irritative symptoms (frequency, urgency, nocturia). It is important to note that LUTS can result from a variety of conditions including problems relating to bladder innervation and aging as well as the outflow obstruction caused by BPH. LUTS due to BPH increases with age, BPH was primarily treated surgically for many years, however, in the 1990s this was superseded by the medical approaches that are now the front line therapy. 5α-reductase inhibitors such as finasteride and dutasteride and α-adrenergic blockers such as doxazosin and tamsulosin are used to shrink and relax the organ, respectively. The MTOPS study demonstrated that a combination of the α-blocker Doxazosin and the 5α-reductase inhibitor Finasteride are more effective at reducing LUTS progression than either drug given alone. While these approaches are effective in many patients, a significant proportion, in the range of 35%, showed progressive disease even in the face of the two drug combination,The Electromagnetic field is thought to have the ability to affect the cells that induce different cellular changes , present studies prove that molecular synergies may not remain the unique determinants implicated in the biological interface. EMF possesses numerous well-reported biological effects including inflammation and pain suppression. This therapy is noninvasive, secure, and easy to use for treating the origin of discomfort, damage, and inflammation

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a condition in which the prostate gland grows larger than normal, but the growth is not caused by cancer .The prostate has two main growth phases. The first growth phase happens early in puberty when the prostate doubles in size. The second growth phase starts around age 25 and continues throughout life. BPH often occurs late in the second growth phase Experts estimate that BPH affects 5% to 6% of men ages 40 to 64 and 29% to 33% of those ages 65 and older. BPH is the most common prostate problem in men older than age 50. BPH rarely causes symptoms in men younger than age 40,Benign prostatic hyperplasia (BPH) is a prostate volume (PV) enlargement due to a non-malignant cellular proliferation of the parenchyma and stroma of the gland, mainly in the transition area. BPH is a common age-related pathology, often causing lower urinary tract symptoms (LUTS) due to compression of the urethra by the enlarged prostate, which reduces the quality of life of affected patients , Pulsed electromagnetic field (PEMF) appears to act on BPH through anti-inflammatory and microvascular effects that can translate into symptomatic improvement. Experimental and translational work suggests PEMF improves prostate microcirculation and reduces tissue inflammation markers, which may decrease stromal/epithelial hyperplasia and interstitial edema-mechanisms that plausibly reduce prostate volume and obstructive lower urinary tract symptoms (LUTS). This proposed mechanism is supported by Doppler/ultrasound findings and physiologic measures reported in preclinical and human pilot studies showing improved prostatic blood flow and reduced inflammatory indices after PEMF treatment ,Regular physical exercise has been shown to positively influence benign prostatic hyperplasia (BPH), a common condition in aging men characterized by prostate enlargement and lower urinary tract symptoms (LUTS). The mechanisms by which exercise may improve BPH including hormonal modulation through reducing insulin-like growth factor-1 (IGF-1) and estrogen levels, both of which are linked to prostate growth, while increasing testosterone metabolism, potentially slowing BPH progression Physical activity (PA) has myriad health benefits, which may also extend to protection against BPH and LUTS development and progression. PA has been proposed to protect against BPH/LUTS by several possible mechanisms, including reducing body size, decreasing sympathetic nervous system activity ,The complications of benign prostatic hyperplasia may include: acute urinary retention, chronic, urinary retention, blood in the urine, urinary tract infections (UTIs), bladder damage and kidney damage Pulsed electromagnetic field therapy (PEMF) consists of low-frequency pulsed energy waves (1-50) Hz, that have been employed for many therapeutic purposes mainly because of its anti-inflammatory effect Moreover, many studies have shown that it is a safe procedure, without side effects ,Emerging evidence demonstrates that regular physical activity significantly enhances quality of life for men with benign prostatic hyperplasia (BPH). found that moderate-intensity aerobic exercise (30-60 minutes, 3-5 times weekly) improved International Prostate Symptom Score (IPSS) by an average of 3.2 points and quality of life scores by 1.5 points compared to sedentary controls. The study attributed these benefits to reduced prostatic inflammation and improved pelvic floor muscle function ,Human observational studies and reviews support that higher levels of physical activity-including aerobic modalities-are associated with lower odds of BPH and LUTS. A systematic review and meta analysis of observational studies found that compared to sedentary lifestyle, moderate to vigorous physical activity was linked to a significantly reduced risk of BPH/LUTS. While randomized controlled evidence remains limited and rated as very low certainty, some small trials (including tai chi and pelvic floor training) demonstrated improvements in symptom scores (e.g. IPSS reduction by ~6-8 points) when compared to waiting or conventional treatment. Together, these findings suggest that regular aerobic exercise may reduce urinary frequency, nocturia, urgency, and weak urinary stream associated with BPH, possibly via metabolic and anti inflammatory mechanisms ,The present study aimed to evaluate the comparative effects of pulsed electromagnetic field (PEMF) therapy and aerobic exercise training on prostatic function in elderly males diagnosed with benign prostatic hyperplasia (BPH). Seventy-five participants were randomly assigned into three equal groups: Group (A) received EMF therapy in addition to medical treatment program, Group (B) received aerobic exercise training in addition to medical treatment program, and Group (C) received medical treatment program alone. Baseline characteristics, including age and body mass index (BMI), revealed no statistically significant differences among the three groups, confirming their initial comparability. Following the intervention period, all groups demonstrated significant within-group improvements in clinical measures, including prostate volume, serum prostate-specific antigen (PSA), the International Prostate Symptom Score (IPSS), the American Urological Association Symptom Index (AUA-SI), and the Older People's Quality of Life Questionnaire (OPQOL-35). However, the extent of improvement varied across the groups,All groups showed significant improvements in prostate volume, PSA, IPSS, AUA-SI, and OPQOL-35 scores. However, Group (A) (PEMF) showed the most notable improvements, particularly in symptom scores and quality of life. These outcomes suggested that PEMF therapy may improve prostatic health by reducing inflammation, enhancing vascular function, and modulating cellular activity.

The findings aligned with emerging literature supporting PEMF's regenerative and anti-inflammatory effects, though its application in urology remains underexplored. This study provided promising evidence for incorporating PEMF therapy into physiotherapy for BPH, offering a safe, effective, and well-tolerated alternative to invasive management for elderly patients, This study provided strong evidence supporting that pulsed electromagnetic field (PEMF) therapy as an effective, non-invasive adjunct for managing Benign Prostatic Hyperplasia (BPH) in elderly men. PEMF improved both objective outcomes, such as prostate volume, and subjective measures, including LUTS and quality of life, without the adverse effects often associated with pharmacological or surgical treatments.

ELIGIBILITY:
Inclusion Criteria:

* Seventy five male elderly patients diagnosed with prostatic enlargement (prostate volume is greater than 40 mL) assessed by ultrasonography.
* They had benign prostatic hyperplasia indicated by a serum-based prostate-specific antigen (PSA) of 4.0 - 10 ng/mL
* They had moderate severity of benign prostatic hyperplasia indicated by a score of 8 to 19 according to the American Urological Association Symptom Index.
* They had lower urinary tract symptoms including nocturia, incomplete emptying of the bladder, urinary hesitancy, weak stream, frequency, and urgency leading to the development of acute urinary retention.

Exclusion Criteria:

* Previous prostatic surgery.
* Urogenital malformations, genetic syndromes, and ongoing tumors.
* Uncontrolled hypertension
* Pacemakers and automatic implantable cardioverter defibrillators.
* Neurological disorders such as Parkinson's disease.
* Prostate cancer.
* Patients taking medications that affected bladder function such as antihistamines, decongestants, diuretics, opiates, and tricyclic antidepressants.

Ages: 60 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only male participants because of our study on volume prostate
Enrollment: 75 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
prostate volume | after 12 weeks of treatment
  This procedure required little to no special preparation, comfortable clothing. The patient was asked to wear a gown and to lie on his side with his knees toward his chest. To obtain high-quality images, an ultrasound transducer - a plastic cylinder about the size of a finger - was inserted a short distance into the rectum. The transducer was covered with a protective sheath and lubricated with gel.

SECONDARY OUTCOMES:
International prostate symptom score (IPSS) | after 12 weeks of treatmen
  There are 7 questions relating to different symptoms the patient may be experiencing and one question relating to his overall quality of life. Once the patient scored each question, the values were added together to give an indication of the severity of the patient symptoms,The score is graded as 0-7: Mild 8-19: Moderate 20-35: Severe
The Older People's Quality of Life Questionnaire (OPQOL-35) | after 12 weeks of treatment
  contains 35 items tapping into eight domains including life overall, health, social relationships and participation, independence, control over life and freedom, home and neighborhood, psychological and emotional well-being, financial circumstances, culture and religion. The participant was asked to indicate the extent to which agreed with every single statement by choosing one of five possible options among "strongly disagree", "disagree", "neither agree nor disagree", "agree" and "strongly agree"

CONTACTS AND LOCATIONS:
Overall Officials: El-Sayed Essam, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo, El Mohandsen, Egypt

IPD SHARING:
Plan to Share IPD: No
because of its indivdual data